CLINICAL TRIAL: NCT00977054
Title: Double Filtration Plasmapheresis (DFPP) in Combination With Pegylated Interferon Alfa-2a and Ribavirin for Patients With Chronic Hepatitis C With Genotype 1 and High Viral Load: a Randomized Controlled Trial
Brief Title: Double Filtration Plasmapheresis for Hepatitis C Virus (HCV) Genotype 1 Patients With High Viral Load
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Novel HCV DAA approved by FDA
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200904053D
Record Dates: First submitted 2009-09-13; First posted 2009-09-15 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Peginterferon alfa-2a; Ribavirin; Plasmapheresis; Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFPP and Peg-IFN + RBV (Experimental): Double filtration plasmapheresis (Day 1, Day 2, Day 4, Day 8, and Day 9 from the onset of treatment; overall 5 session, each session for 4 hours) and weekly subcutaneous peginterferon alfa-2a 180 ug (week 1 to week 48) and daily oral ribavirin 1,000-1,200 mg (week 1 to week 48; body weight < 75 kg, 1,000 mg/day and body weight >= 75 kg, 1,200 mg/day)
  Interventions: Drug: DFPP + Peg-IFN + RBV
- Peg-IFN + RBV (Active Comparator): Weekly subcutaneous peginterferon alfa-2a 180 ug (week 1 to week 48) and daily oral ribavirin 1,000-1,200 mg (week 1-48; body weight < 75 kg, 1,000 mg/day and body weight >=75 kg, 1,200 mg/day)
  Interventions: Drug: Peg-IFN + RBV

INTERVENTIONS:
Drug: DFPP + Peg-IFN + RBV — Double filtration plasmapheresis: day 1,2,4,8,9 from the onset of treatment (4 hours for each session) Peginterferon alfa-2a: week 1-48, weekly subcutaneous 180 ug Ribavirin: week 1-48, daily oral 1,000-1,200 mg (body weight < 75 kg, 1,000 mg/day; body weight loss >= 75 kg, 1,200 mg/day)
  Other Names: DFPP: Plasmaflo + Cascadeflo EC-50W (Asahi); Peg-IFN alfa-2a: Pegasys (Hoffman La-Roche); RBV: Copegus (Hoffman La-Roche)
  Arms: DFPP and Peg-IFN + RBV
Drug: Peg-IFN + RBV — Peginterferon alfa-2a: week 1-48, weekly subcutaneous 180 ug Ribavirin: week 1-48, daily oral 1,000-1,200 mg (body weight < 75 kg, 1,000 mg/day; body weight loss >= 75 kg, 1,200 mg/day)
  Other Names: Peg-IFN alfa-2a: Pegasys (Hoffman La-Roche); RBV: Copegus (Hoffman La-Roche)
  Arms: Peg-IFN + RBV

SUMMARY:
Hepatitis C virus (HCV) infection, a leading cause of cirrhosis, hepatocellular carcinoma (HCC) and liver transplantation, affects approximately 170 million individuals worldwide. The prevention of HCV transmission and early intervention of HCV infection are urgently needed to reduce or halt the liver-related morbidity and mortality. Double filtration plasmapheresis (DFPP) has been with widespread use in clinical practice for several indications with plasma filters optimized for the respective elimination targets with excellent safety. By way of the plasma separator, the blood is separated into plasma and cell components. Separated plasma is then led into the plasma component separator where the pores of the plasma component separator further fractionate the plasma into large and small molecular components. The large molecular components, including pathogenic substances, is removed and discarded and the small molecular components, including proteins such as albumin and gamma-globulin, are returned to the patient and mixed with the cell components. After the initiation of pegylated interferon plus ribavirin (Peg-IFN+RBV) therapy, the rapid first phase relates to a significant reduction in virus production and the degradation of free virus particles, which is followed by a second much slower one reflecting the elimination and clearance of infected cells. In HCV patients, high baseline viral load at the initiation of therapy is considered to be a negative predictor for systemic vascular resistance (SVR) for HCV genotype 1 patients. Reduction of baseline viral load by means of therapeutic double filtration plasmapheresis (DFPP) may represent a plausible adjunct for improved antiviral therapy to reduce the virus load with the initiation of treatment in synergy with Peg-IFN and RBV combination therapy. Recently, several clinical studies in evaluating the therapeutic efficacy and safety of DFPP in conjunction with IFN-based therapy were conducted for treatment-naïve genotype 1 high viral load CHC patients, and CHC patients who underwent liver transplantation. These studies showed that patients with DFPP treatment had more favorable HCV early viral kinetics to those without DFPP treatment. Furthermore, all these studies showed excellent safety after DFPP treatment. Therefore, the investigators aimed to conduct a large-scaled randomized controlled trial to evaluate the overall response of DFPP for HCV genotype 1 patients with high viral load.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection, a leading cause of cirrhosis, hepatocellular carcinoma (HCC) and liver transplantation, affects approximately 170 million individuals worldwide. The prevention of HCV transmission and early intervention of HCV infection are urgently needed to reduce or halt the liver-related morbidity and mortality. Currently, combination therapy with peginterferon (Peg-IFN) and ribavirin (RBV) has become the standard of care for chronic hepatitis C (CHC) patients, with an overall sustained virologic response (SVR) rate of 54-63%. Treatment with weekly Peg-IFN and weight-based RBV for 48 weeks resulted in a significantly higher SVR rate than that for 24 weeks in patients with HCV genotype 1 infection. While HCV genotype 1 patients who had both rapid virologic response (RVR) and low pretreatment viral load could receive short duration of therapy without compromising the treatment responses, those who had either high baseline viral load or failed to achieve RVR should receive at least 48 weeks of treatment. RVR is considered the most important factor for SVR. Furthermore, several studies have repeated shown that high baseline viral load (> 400,000~800,000 IU/mL) was closely associated with failure to achieve RVR in these patients. Therefore, efforts to improve the RVR rate is important to facilitate the overall treatment responses.

Double filtration plasmapheresis (DFPP), a well established method of therapeutic apheresis, has been with widespread use in clinical practice for several indications with plasma filters optimized for the respective elimination targets. By way of the plasma separator, the blood is separated into plasma and cell components. Separated plasma is then led into the plasma component separator where the pores of the plasma component separator further fractionate the plasma into large and small molecular components. The large molecular components, including pathogenic substances, is removed and discarded and the small molecular components, including proteins such as albumin and gamma-globulin, are returned to the patient and mixed with the cell components.

DFPP has been used in the treatment of many diseases such as neurological diseases, collagen diseases, hematological diseases, skin diseases, and renal diseases, and its efficacy and safety have been well established. It is noteworthy to mention that DFPP has been indicated to treat CHC in Japan since April 2008. In Germany, the safety of DFPP in LDL-apheresis was analyzed within a retrospective multicenter investigation including data from 1702 ambulatory DFPP-LDL-apheresis treatments of 52 patients (REMUKAST Study). Ninety-eight percent of the treatments bear no serious adverse events while only 2% of slight hypotensive episodes were observed. In a recent investigation, efficacy and safety of DFPP was compared with the HELP (Heparin-induced Extracorporeal LDL-Cholesterol Precipitation) system in a cross-over design. No serious adverse events occurred in this study including 44 treatments.

During chronic infection, the level of serum HCV RNA is in a steady state with only minor fluctuations in untreated patients. A dynamic equilibrium, involving hepatocytes and plasma components, exists between new viral production and viral destruction during chronic HCV infection. After the initiation of Peg-IFN plus RBV therapy, the viral decline can be divided into two major phases. Over the first 24 - 48 h the initial dose of PEG-IFN/RBV leads to a first decline of HCV RNA which ranges from 0.5-2.0 log levels. This rapid first phase relates to a significant reduction in virus production and the degradation of free virus particles, which is followed by a second much slower one reflecting the elimination and clearance of infected cells.

As described above, a high baseline viral load (HCV-RNA > 800,000 IU/mL) at the initiation of therapy is considered to be a negative predictor for SVR for HCV genotype 1 patients. Reduction of baseline viral load by means of therapeutic DFPP may represent a plausible adjunct for improved antiviral therapy to reduce the virus load with the initiation of treatment in synergy with Peg-IFN and RBV combination therapy. Therefore the rationale for the effect of DFPP is that the reduced amount of virus during the initiation phase supports the therapeutic efficacy of Peg-IFN and RBV combination therapy by preventing liver reinfection by circulating HCV.

Recently, several small-scaled clinical studies in evaluating the therapeutic efficacy and safety of DFPP in conjunction with IFN-based therapy were conducted for treatment-naïve genotyp1 high viral load CHC patients, and CHC patients who underwent liver transplantation. These studies showed that patients with DFPP treatment had more favorable HCV early viral kinetics to those without DFPP treatment. The large-scaled non-randomized clinical study totally evaluating 104 CHC patients showed that the addition of DFPP had a higher SVR rate to those without DFPP treatment in HCV genotype 1 patients with baseline viral load > 100,000 IU/mL (70.8% versus 50.0%), probably due to eliminating a substantial part of viral particles from the dynamic equilibrium of the liver and plasma compartments. Furthermore, all these studies showed excellent safety after DFPP treatment. However, these studies were limited by the small case numbers and non-randomized assignment, making the role of DFPP in improving the efficacy of difficult-to-treat HCV patients still debated. Therefore, the investigators aimed to conduct a large-scaled randomized controlled trial to evaluate the overall response of DFPP for HCV genotype 1 patients with high viral load.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve
* Age 18 and older
* Anti-HCV (Abbott HCV EIA 2.0, Abbott Diagnostic, Chicago, IL) positive > 6 months
* Detectable serum quantitative HCV-RNA (Cobas Taqman v2.0, Roche Diagnostics) with HCV RNA > 800,000 IU/mL
* HCV genotype 1 (Inno-LiPA, Innogenetics)
* A liver biopsy consistent with the diagnosis of chronic hepatitis C

Exclusion Criteria:

* Anemia (hemoglobin < 13 gram per deciliter for men and < 12 gram per deciliter for women)
* Neutropenia (neutrophil count <1,500 per cubic milliliter)
* Thrombocytopenia (platelet <90,000 per cubic milliliter)
* Co-infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Chronic alcohol abuse (daily consumption > 20 gram per day)
* Decompensated liver disease (Child-Pugh class B or C)
* Serum creatinine level more than 1.5 times the upper limit of normal
* Autoimmune liver disease
* Neoplastic disease
* An organ transplant
* Immunosuppressive therapy
* Poorly controlled autoimmune diseases, pulmonary diseases, cardiac diseases, psychiatric diseases, neurological diseases, diabetes mellitus
* Evidence of drug abuse
* Unwilling to have contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | 18 months

SECONDARY OUTCOMES:
Rapid virologic response (RVR) | 1 month
Treatment-related withdrawal rate | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Study Chair — National Taiwan University Hospital; Jia-Horng Kao, MD, PhD, Study Director — National Taiwan University Hospital; Shih-Jer Hsu, MD, Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch; Cheng-Chao Liang, MD, BS, Principal Investigator — Far Eastern Memorial Hospital; Hung-Bin Tsai, MD, Principal Investigator — Buddhist Tzu Chi General Hospital; Peir-Haur Hung, MD, Principal Investigator — Chiayi Christian Hospital; Chih-Lin Lin, MD, BS, Principal Investigator — Taipei Municipal Hospital, Ren-Ai Branch
Locations (6):
- Taiwan (6):
  - Buddhist Tzu Chi General Hospital, Chiayi City
  - Chiayi Christian Hospital, Chiayi City
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - Far Eastern Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Municipal Hospital, Taipei